CLINICAL TRIAL: NCT04579991
Title: Effects of Visnadin, Ethyl Ximeninate, Coleus Barbatus and Millet in Emulgel on Sexual Function in Postmenopausal Women With Vulvovaginal Atrophy, a Randomized Controlled Trial
Brief Title: Effects of Visnadin, Ethyl Ximeninate, Coleus Barbatus and Millet in Emulgel on Sexual Function in Postmenopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRU20200001
Record Dates: First submitted 2020-10-06; First posted 2020-10-08 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Female Sexual Function; Vulvovaginal Atrophy; Postmenopausal Atrophic Vaginitis
Keywords: Vulvovaginal atrophy; Genitourinary Syndrome of Menopause; Postmenopausal women; Female sexual function; Visnadin
MeSH Terms: conditions — Atrophic Vaginitis | interventions — visnadin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacist will provide the same color and texture of product and identical package for both active emulgel and emulgel only products. She is the only person who knows the code of product and prepare the product in the opaque envelop for all participants.
  The statistician will generate the code of product to all participants with block-of-four randomization method.
  The nurse will distribute and help the participants fill all questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Active Comparator): Apply small amount of topical visnadin, ethyl ximeninate, coleus barbatus and millet in emulgel on mucosal surface of vulva included clitoris every day before bedtime for 8-week period.
  Interventions: Other: Visnadin, ethyl ximeninate, coleus barbatus and millet in emulgel
- Placebo Group (Placebo Comparator): Apply small amount of topical emulgel-only on mucosal surface of vulva included clitoris every day before bedtime for 8-week period.
  Interventions: Other: Emulgel-only

INTERVENTIONS:
Other: Visnadin, ethyl ximeninate, coleus barbatus and millet in emulgel — Topical product, apply small amount on mucosal surface of vulva included clitoris once daily
  Arms: Active Group
Other: Emulgel-only — Topical placebo product, apply small amount on mucosal surface of vulva included clitoris once daily
  Arms: Placebo Group

SUMMARY:
This clinical trial, a double blind randomized controlled trial, is conducted to determine the effects of daily topical visnadin, ethyl ximeninate, coleus barbatus and millet in emulgel on sexual function in postmenopausal women with vulvovaginal atrophy within 8-week of treatment. We compare the active ingredient in emulgel to the emulgel only. We also evaluate the improvement of the vulvovaginal atrophy symptoms in postmenopausal women, the safety and the tolerability of visnadin, ethyl ximeninate, coleus barbatus and millet in emulgel. This study is conducted in the Menopause Clinic and the Gynecology Clinic, King Chulalongkorn Memorial Hospital, Bangkok, Thailand.

DETAILED DESCRIPTION:
Topical visnadin, ethyl ximeninate, coleus barbatus and millet in emulgel is a cosmetic product. Visnadin is an active ingredient which has the vasodilator effect and improve blood flow to female vulvovaginal area. This will improve lubrication from increase Bartholin's gland secretion. As the clitoral blood flow increase, the sexual response could be improved. The ethyl ximeninate, coleus barbatus and millet are plant extract which have moisturizer, anti-inflammation and antioxidant effects. Our hypothesis is a daily topical visnadin, ethyl ximeninate, coleus barbatus and millet in emulgel could improved sexual function and vulvovaginal atrophic symptoms in postmenopausal women with vulvovaginal atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Women age 45-65 years old
* BMI 19-29 kg/m2
* Menopause or removal of both ovaries more than 1 year
* Has moderate to severe vulvovaginal atrophic at least 1 symptom
* Has sign of vulvovaginal atrophy
* Vaginal pH ≥ 5
* Has sexual intercourse at least 1 time/month

Exclusion Criteria:

* Hormonal use within 3 months
* Use vaginal estrogen/ moisturizer within 3 months
* Use aromatase inhibitor/tamoxifen within 3 months
* Has vaginal bleeding within 6 months
* Acute or chronic urinary tract infection
* History of radiation therapy at vulvovaginal and pelvic area
* History of Diabetes mellitus or Cardiovascular disease
* History of neurosis or psychosis
* History of vulvovaginal cancer
* History of smoking more than 20 cigarettes/day
* History of alcoholic drink/ drug abuse
* History of visnadin, ethyl ximeninate, coleus barbatus and millet allergy
* Has disease of vulva

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 100 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-11-25 (Estimated)

PRIMARY OUTCOMES:
Sexual function | 8-week
  Female Sexual Function Index (FSFI) The full scale (overall) score of the FSFI can be derived from the six domain scores; desire, arousal, lubrication, orgasm, satisfaction and pain. The minimum value is 2.0 and maximum value is 36.0, and the higher scores mean a better outcome.
Vulvovaginal atrophic symptoms score | 8-week
  4-likert scale; 0 = no symptom, 1= mild symptom, 2 = moderate symptom, 3 = severe symptom The minimum is 0 and maximum value is 4, and the higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Adverse event and tolerability | 8-week
  Possible adverse event of therapeutic use

CONTACTS AND LOCATIONS:
Overall Officials: Sukanya Chaikittisilpa, MD,MSc, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No